CLINICAL TRIAL: NCT06207110
Title: Addressing Appetitive Traits to Promote Weight Management in Children Who Overeat
Brief Title: Family, Responsibility, Education, Support, and Health for Food Responsiveness
Acronym: FRESH-FR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Minnesota (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kerri Boutelle, Kerri Boutelle, Ph.D.,, Professor of Pediatrics, Psychiatry, and Herbert Wertheim School of Public Health and Human Longevity Science, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 806055; 1R01DK135599 (NIH)
Record Dates: First submitted 2024-01-05; First posted 2024-01-16 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Obesity, Childhood
Keywords: Food Responsiveness; Satiety Responsiveness; Weight Loss; Overeating
MeSH Terms: conditions — Pediatric Obesity; Weight Loss; Hyperphagia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Regulation of Cues (Experimental): The ROC program provides psychoeducation, coping skills, self-monitoring and experiential learning targeting increasing satiety responsiveness and decreasing food cue responsiveness.
  Interventions: Behavioral: Regulation of Cues
- Family-Based Treatment (Active Comparator): The FBT program provides nutrition and physical activity education, behavior therapy skills, and parenting skills targeting changes in energy balance.
  Interventions: Behavioral: Family Based Behavioral Treatment
- Regulation of Cues + (Experimental): The ROC+ program includes all of the components of ROC as well as nutrition education and reducing energy intake
  Interventions: Behavioral: Regulation of Cues +
- Health Education (Active Comparator): The HE program provides information about nutrition, physical activity, sedentary behavior, sleep, emotions, and stress.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Regulation of Cues — ROC is based on the Behavioral Susceptibility Theory and designed to incorporate psychoeducation, cue-exposure treatment, appetite awareness training, coping skills, and self-monitoring of satiety and cravings to improve satiety responsiveness and decrease food cue responsiveness. This arm will include an experiential component, including hunger monitoring during a meal or snack and participating in exposure exercises.
  Other Names: ROC
  Arms: Regulation of Cues
Behavioral: Family Based Behavioral Treatment — FBT provides nutrition and physical activity education, behavior therapy skills, and parenting skills targeting changes in energy balance.
  Other Names: FBT
  Arms: Family-Based Treatment
Behavioral: Regulation of Cues + — ROC+ includes all of the skills provided in ROC but integrates nutrition education and reducing energy intake
  Other Names: ROC+
  Arms: Regulation of Cues +
Behavioral: Health Education — The HE program provides information about nutrition, physical activity, sedentary behavior, sleep, emotions, and stress.
  Other Names: HE
  Arms: Health Education

SUMMARY:
The objective of this proposed study is to compare Regulation of Cues (ROC), Family-Based Treatment (FBT), ROC+ nutrition education and reducing energy intake (ROC+) and a health education comparator (HE) for children with overweight or obesity who are high on food responsiveness (FR).

DETAILED DESCRIPTION:
The investigators have developed a new model for the treatment of obesity, called Regulation of Cues (ROC), which is based on Behavioral Susceptibility Theory. The ROC program targets two theorized mechanisms for overeating; decreased sensitivity to appetitive cues and increased sensitivity to external food cues. Considering that FBT has merit for some children, but not all, this study will compare ROC to FBT, ROC with nutrition education and reducing energy intake (ROC+), and Health Education (HE). Treatment will consist of weekly individual sessions for the first 16 sessions, then twice per month for the final 2 months for a total of 20 sessions. The investigators will recruit children ages 7-12 with overweight or obesity who are high in food responsiveness (FR) and their parent and will conduct assessments at baseline, post-treatment (month 6), 6-month follow-up (month 12) and 12-month follow-up (month 18).

ELIGIBILITY:
Inclusion Criteria:

1. Informed assent and parental consent
2. A child with overweight or obesity (≥ 85th BMI%) aged 7-12 years of age
3. Child high on FR - High FR will be measured by the Food Responsiveness Scale via the CEBQ, with scores at a 3.8 or higher constituting a child with high FR.
4. A parent responsible for food preparation who is willing to participate and can read, speak and understand English at a minimum of a 5th grade level
5. Family is willing to commit to attending all assessment and treatment sessions, agree to be randomized and participate in all aspects of potential treatments
6. Child is on stable medication regimen for medications that can impact weight (3+ months)
7. Child does not have medical conditions that limit ability to participate in physical activity for the duration of the study. Parent can participate in physical activity with their child or provide opportunities for the child to complete recommended physical activity

Exclusion Criteria:

1. Acute child psychiatric disorder diagnoses (e.g., acute suicidality, recent hospitalization, psychosis, bulimia nervosa)
2. Child diagnoses of a serious chronic physical disease (e.g., cystic fibrosis, type 1 diabetes) for which physician supervision of diet and exercise prescription may be warranted
3. Child who is taking medication for weight loss
4. Acute parent psychiatric disorder (e.g., acute suicidality; recent hospitalization; psychosis, bipolar disorder, borderline personality disorder, moderate or severe alcohol or substance use disorder)
5. First degree relative or someone in the household with anorexia or bulimia nervosa.

Potential participants with medical or psychological diagnosis that could make adherence with the study protocol difficult or dangerous will not be included.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Child age and sex adjusted body mass index z-score (BMIz) | Change from baseline at 3 months, 6 months, 12 months, and 18 months
  Age and sex adjusted body mass index (BMI (kg/m^2)) z-score based on the Centers for for Disease Control and Prevention (CDC) norms
Child percentage of the 95th percentile BMI (%BMIp95) | Change from baseline 3 months, 6 months, 12 months, and 18 months
  Age and Sex specific percentage of the 95th percentile BMI
Change in Child Overeating | Change from baseline at 6 months,12 months, and 18 months
  Measured by The Eating in the Absence of Hunger Questionnaire; Scores ranging from 1-5 with greater scores meaning more eating in the absence of hunger.

SECONDARY OUTCOMES:
Child Food Cue Responsiveness as measured by the Child Eating Behavior Questionnaire | Change from baseline at 6 months,12 months, and 18 months]
  The Food Responsiveness (FR) Scale of the Child Eating Behavior Questionnaire; scores range from 1-5 with higher scores representing greater FR.
Child Food Cue Responsiveness as measured during exposure to a preferred food | Change from baseline at 6 months,12 months, and 18 months
  The child will be asked to hold, smell, and taste the highly craved food and rate their current cravings over the course of 5 minutes.
Child Satiety Responsiveness as measured by the Child Eating Behavior Questionnaire | Change from baseline at 6 months,12 months, and 18 months
  The Satiety Responsiveness (SR) scale of the Child Eating Behavior Questionnaire (CEBQ). Scores range from 1-5 with higher scores representing greater SR.
Child Satiety Responsiveness as measured by the Water Load Task (WLT) | Change from baseline at 6 months,12 months, and 18 months
  The Water Load Task
Child Inhibition as measured by the Stop Signal Task | Change from baseline at 6 months,12 months, and 18 months
  Stop Signal Task with food stimuli
Child Inhibition as measured by the Go No Go (GNG) Task | Change from baseline at 6 months,12 months, and 18 months
  The Go No Go (GNG) task with food stimuli
Child Energy Intake | Change from baseline at 6 months,12 months, and 18 months
  Automated Self-Administered 24-hour recall (ASA-24)
Parent Body Mass Index (BMI) | Change from baseline at 3 months, 6 months,12 months, and 18 months
  kg/m^2
Parent Overeating | Change from baseline at 6 months,12 months, and 18 months
  Eating in the Absence of Hunger Questionnaire; Scores ranging from 1-5 with greater scores meaning more eating in the absence of hunger.
Parent Food Cue Responsiveness as measured by the Adult Eating Behavior Questionnaire | Change from baseline at 6 months,12 months, and 18 months
  Measured by the Food Responsiveness (FR) Scale of the Adult Eating Behavior Questionnaire (AEBQ); scores range from 1-5 with higher scores equating to higher FR.
Parent Food Cue Responsiveness as measured during exposure to a preferred food | Change from baseline at 6 months,12 months, and 18 months]
  The parent will be asked to hold, smell, and taste the highly craved food and rate their current cravings over the course of 5 minutes.
Parent Satiety Responsiveness as measured by the Adult Eating Behavior Questionnaire | Change from baseline at 6 months,12 months, and 18 months
  The Satiety Responsiveness Scale of the AEBQ; scores range from 1-5 with higher scores equating to higher SR
Parent Satiety Responsiveness as measured by the Water Load Task | Change from baseline at 6 months,12 months, and 18 months
  The Water Load Task
Parent Inhibition as measured by the Stop Signal Task | Change from baseline at 6 months,12 months, and 18 months
  Stop Signal Task with food stimuli
Parent Inhibition as measured by the Go No Go (GNG) Task | Change from baseline at 6 months,12 months, and 18 months
  The Go No Go (GNG) task with food stimuli.
Parent Energy Intake | Change from baseline at 6 months,12 months, and 18 months
  Automated Self-Administered 24-hour recall (ASA-24)

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, Ph.D., Principal Investigator — UC San Diego
Locations (2):
- United States (2):
  - UC San Diego Center for Healthy Eating and Activity Research (CHEAR), La Jolla, California
  - Ambulatory Research Center - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more on our study webpage — https://chear.ucsd.edu/research-studies/current-studies